CLINICAL TRIAL: NCT02709863
Title: Comparison of The Effects of Sevoflurane, Desflurane and Total Intravenous Anaesthesia on Pulmonary Function Tests in Patients Undergoing Endoscopic Endonasal Transsphenoidal Surgery of Pituitary Gland
Brief Title: Comparison of The Effects of Sevoflurane, Desflurane and Total Intravenous Anaesthesia on Pulmonary Function Tests
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Abdulvahap Oguz, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 83045809/604.01/02
Record Dates: First submitted 2016-02-23; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Sevoflurane; Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevoflurane (Active Comparator): 1-1.5 minimum alveolar concentration (MAC), inhalation route, during operation
  Interventions: Drug: Sevoflurane
- Desflurane (Active Comparator): 1-1.5 minimum alveolar concentration (MAC), inhalation route, during operation
  Interventions: Drug: Desflurane
- Propofol (Active Comparator): 6-10 mg/kg/h, iv infusion, during operation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — 1-1.5 MAC, inhalation route, during operation
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Desflurane — 1-1.5 MAC, inhalation route, during operation
  Other Names: Suprane
  Arms: Desflurane
Drug: Propofol — 6-10 mg/kg/h, iv infusion, during operation
  Arms: Propofol

SUMMARY:
This study will compare the effects of sevoflurane, desflurane and total intravenous anaesthesia on pulmonary function tests in patients undergoing endoscopic endonasal transsphenoidal surgery of pituitary gland. Participants will be divided into three equal groups. The first group will receive sevoflurane, second grup will receive desflurane and third grup will receive total intravenous anaesthesia. Investigators are also going to evaluate blood gas analysis.

DETAILED DESCRIPTION:
Investigators are going to evaluate forced expiratory volume in 1st Second (FEV1), forced vital capacity (FVC), FEV1/FVC ratio, partial pressure of arterial oxygen (PaO2), partial pressure of arterial carbon dioxide (PaCO2), potential of hydrogen (pH), arterial oxygen saturation (SaO2), base excess (BE), bicarbonate (HCO3) and partial pressure of arterial oxygen/fraction of inspired oxygen (PaO2/FiO2) ratio to compare the effects of drugs.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score I-II patients

Exclusion Criteria:

* Significant cardiopulmonary disease,
* Diagnosed obstructive or restrictive pulmonary disease,
* Patients with chest wall deformities, liver or kidney failure,
* Postoperative lack of cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline FEV1%predicted (no unit) | Preoperative baseline, postoperative 1st hour and postoperative 24th hour
  FEV1 is measured with spirolab III colour liquid-crystal-display medical spirometer. FEV1%predicted is calculated with age, sex, height and weight input by the same equipment.

SECONDARY OUTCOMES:
Change from baseline FVC%predicted (no unit) | Preoperative baseline, postoperative 1st hour and postoperative 24th hour
  FVC is measured with spirolab III colour liquid-crystal-display medical spirometer. FVC%predicted is calculated with age, sex, height and weight input by the same equipment.
Change from baseline FEV1/FVC ratio (no units) | Preoperative baseline, postoperative 1st hour and postoperative 24th hour
  FEV1/FVC ratio is calculated by spirolab III colour liquid-crystal-display medical spirometer based on age, sex, height and weight.
Change from baseline PaO2 (mmHg) | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  PaO2 is a component of arterial blood gas analysis done with Cobas B221.
Change from baseline PaCO2 (mmHg) | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  PaCO2 is a component of arterial blood gas analysis done with Cobas B221.
Change from baseline pH | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  pH is a component of arterial blood gas analysis done with Cobas B221
Change from baseline SaO2 (%) | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  SaO2 is a component of arterial blood gas analysis done with Cobas B221
Change from baseline BE (mmol/L) | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  BE is a component of arterial blood gas analysis done with Cobas B221
Change from baseline HCO3 (mmol/L) | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  HCO3 is a component of arterial blood gas analysis done with Cobas B221
Change from baseline PaO2/FiO2 ratio (no units) | Preoperative baseline, during the 1st hour of the operation, during the last hour of the operation, postoperative 1st hour and postoperative 24th hour
  PaO2/FiO2 ratio is calculated by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Korkmaz Dilmen, Assoc. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty Neurosurgery Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No